CLINICAL TRIAL: NCT03216239
Title: Does Colectomy Predispose to Small Intestinal Bacterial (SIBO) and Fungal Overgrowth (SIFO)
Brief Title: SIBO & SIFO After Colectomy
Status: Completed | Type: Observational
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Satish Rao, Professor of Medicine, Director of Neurogastroenterology/Motility, Augusta University
Other Study IDs: 659642
Record Dates: First submitted 2017-07-11; First posted 2017-07-13 (Actual); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Small Intestinal Bacterial Overgrowth; Small Intestinal Fungal Overgrowth; Colectomy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Colectomy Group: Mean age 52.3 years (range:20-85), 82% females, and a mean duration of symptoms of 79.9 months in the colectomy group. The indication for colectomy was constipation (36%), diverticular disease (8%), bowel obstruction (8%), colorectal carcinoma (8%), colon polyps (6%), and other (34%).
- Control Group: Mean age of 49.9 years (range 18-88), 76% females, and mean duration of symptoms 77.6 months,

SUMMARY:
After subtotal colectomy, 40% of patients report abdominal pain, gas and diarrhea, and poor quality of life; whose etiology is unknown. The investigators determined whether small intestinal bacterial (SIBO or fungal overgrowth SIFO) could cause these sympotoms (> 1 year).

ELIGIBILITY:
Inclusion Criteria:

patients who were referred to a specialist motility center over 4 year period with:

* Unexplained gastrointestinal symptoms such as gas, bloating, belching, diarrhea, and abdominal discomfort
* history of colectomy
* patients with no history of colectomy
* patients included who had normal: upper endoscopy, colonoscopy, computerized abdominal tomography scan, and normal hematology, biochemical profiles, tissue transglutaminase antibody, thyroid stimulating hormone, and normal right upper quadrant ultrasound scan.
* patients with glucose breath test and/or duodenal aspirate

Exclusion Criteria:

* patients with upper gut or small bowel surgery
* Patients who were hospitalized or with serious cardiac or pulmonary or neurologic comorbidities
* Patients with intestinal strictures or known intestinal motility disorders such as scleroderma or pseudo-obstruction syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients of the Digestive Health Center over a 4 year period who have been seen by the motility specialists for unexplained gastrointestinal symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-02-24 (Actual); Primary Completion 2016-02-26 (Actual); Study Completion 2016-02-26 (Actual)

PRIMARY OUTCOMES:
Prevalence of SIBO/SIFO | 4-5 years
  Patients with unexplained GI symptoms following colectomy and to compare this with a control group of patients with similar symptoms but without previous colectomy.

SECONDARY OUTCOMES:
Response to treatment with antibiotics and antifungals | 4-5 years
  Secondary aim was to assess the response to treatment with antibiotics and antifungals in colectomy patiens with SIBO/SIFO